CLINICAL TRIAL: NCT02692209
Title: A Multi-Reader Multi-Case Controlled Clinical Trial to Evaluate the Comparative Accuracy of the Fujifilm FFDM Plus DBT Versus FFDM Alone in the Detection of Breast Cancer
Brief Title: A Multi-Reader Multi-Case Pivotal Trial
Status: Completed | Type: Observational
Sponsor: Fujifilm Medical Systems USA, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: FMSU2013-004G
Record Dates: First submitted 2015-12-08; First posted 2016-02-25 (Estimated); Results first posted 2020-06-11 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-06

CONDITIONS: Breast Cancer
Keywords: Mammography
MeSH Terms: conditions — Breast Neoplasms | interventions — Mammography

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- FFDM Plus DBT: FFDM Plus DBT images are being evaluated as compared to FFDM alone
  Interventions: Device: FFDM Plus DBT
- Full Field Digital Mammography: Fujifilm FFDM alone images are being evaluated as compared to FFDM + DBT
  Interventions: Device: FFDM Alone

INTERVENTIONS:
Device: FFDM Plus DBT — FFDM + DBT Images
  FujiFilm Aspire Cristalle System
  Groups: FFDM Plus DBT
Device: FFDM Alone — FFDM Alone Images
  Groups: Full Field Digital Mammography

SUMMARY:
The purpose of this pivotal reader study is to assess the comparative accuracy of Fujifilm FFDM plus DBT versus FFDM alone in the detection of breast cancer.

DETAILED DESCRIPTION:
The safety and effectiveness of FFDM + DBT are both linked to the ability of radiologists interpreting FFDM + DBT images to accurately diagnose breast cancer. Each study endpoint therefore addresses both safety and effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* Eligible subjects under protocol FMSU2013-004A, defined as female subjects with known true clinical status and with complete FFDM and DBT examinations, in which there is sufficient anatomical coverage, sufficient contrast, and no significant motion or other artifacts, as determined by the image-acquisition sites.
* Meet none of the exclusion criteria under protocol FMSU2013-004A.

Exclusion Criteria:

* Subjects who are in violation of protocol FMSU2013-004A.
* Subjects who meet exclusion criteria under protocol FMSU2013-004A.
* Subjects with unknown clinical status.
* Any subject whose positive mammogram was not read during the truthing process (see section 8) will not be considered for the pivotal MRMC reader study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This research is a retrospective study with an enriched sample of breast screening or diagnostic cases that were selected from the library of mammograms collected under Fujifilm protocol FMSU2013-004A.
Sampling Method: Probability Sample
Enrollment: 298 (Actual)
Dates: Start 2015-12; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert M Uzenoff, Study Director — Fujifilm Medical Systems USA, Inc.
Locations (5):
- United States (5):
  - Scottsdale Medical Imaging, Ltd, Scottsdale, Arizona
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Elizabeth Wende Breast Care, LLC (EWBC), Rochester, New York
  - University of North Carolina - at Chapel Hill, Chapel Hill, North Carolina
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The 298 breast screening and diagnostic cases selected for this study, were obtained from the FMSU2013-004A acquisition study. The statistician randomly selected cases to provide a distribution of density, finding types, etc.
Pre-assignment Details: Reading radiologists independently read all 298 cases sequentially; first as an FFDM read, then as a FFDM + DBT read on the Aspire Bellus workstation.
  There was no washout, and all data below is entered correctly.
Groups:
- FFDM Alone Then FFDM Plus DBT: FFDM images are being evaluated as compared to FFDM Plus DBT
  FujiFilm Aspire Cristalle System
  This is a sequential read, each reader read the case as a FFDM read followed by a FFDM plus DBT read
Period: Overall Study
Arm/Group | FFDM Alone Then FFDM Plus DBT
Started | 298
Completed | 298
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: There were 298 study participants in total who had their images reviewed by 28 radiologist readers. Images were acquired under acquisition study FMSU2013-004A.
Groups:
- All 298 Cases/Study Participants: There were 298 study participants in total who had their images reviewed by 28 radiologist readers. Images were acquired under acquisition study FMSU2013-004A.
Arm/Group | All 298 Cases/Study Participants
Number analyzed (Participants) | 298
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 59 [49 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 298
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 23
  White | 269
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 298

OUTCOME MEASURES:

1. Primary Outcome: Correct Lesion Localization: Area Under the Receiver Operating Characteristic (ROC) Curve (AUC) for FFDM + DBT Versus FFDM Alone Based on Probability of Malignancy (POM) Scores and Requiring Correct Lesion Localization.
Description: The study will be considered to have successfully demonstrated safety and effectiveness of the Fujifilm Aspire Cristalle: FFDM +DBT system if the per-subject average AUC for FFDM+DBT is statistically significantly superior to the average AUC for FFDM alone at the alpha = 0.05 significance level. Per-subject BI-RADS, POM and recall scores requiring correct lesion localization were derived. The general principle is that even at the subject level, credit was only given for identifying a subject with cancer if the reader marked findings in at least one location with cancer. When computing sensitivity and specificity based on BI-RADS, a score of 4 or 5 constituted a positive test result.
Time Frame: 1 month
Population: Twenty-eight qualified radiologists independently performed reads on all 298 cases. Each radiologist reader read each case sequentially, first as a FFDM read, and then FFDM + DBT read, all on the Aspire Bellus workstation.
Measure: Mean (95% Confidence Interval); unit: Probability
Groups:
- FFDM Plus DBT: FFDM Plus DBT images are being evaluated as compared to FFDM alone
  FFDM Plus DBT: FFDM + DBT Images
  FujiFilm Aspire Cristalle System
- Full Field Digital Mammography (FFDM): Fujifilm FFDM alone images are being evaluated as compared to FFDM + DBT
  FFDM Alone: FFDM Alone Images
Arm/Group | FFDM Plus DBT | Full Field Digital Mammography (FFDM)
Number analyzed (Participants) | 298 | 298
Probability | 0.837 [0.788 to 0.886] | 0.784 [0.726 to 0.841]

ADVERSE EVENTS:
Time Frame: 5 weeks
Description: There were no AE's expected for this study, as it was a radiologist reader study utilizing retrospective imaging. No study subjects were on-site for this retrospective review. No Adverse Events to report.
Arm/Group | FFDM Plus DBT | Full Field Digital Mammography
All-Cause Mortality (participants affected / at risk) | 0/298 | 0/298
Serious Adverse Events (participants affected / at risk) | 0/298 | 0/298
Other Adverse Events (participants affected / at risk) | 0/298 | 0/298

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No